CLINICAL TRIAL: NCT07170202
Title: Translating Behavioral Economics Strategies to Culturally Tailor a Mobile Health Mindfulness Intervention to Reduce Risky Drinking Behaviors in Black College Student Men
Brief Title: The Increasing Mindfulness Engagement Project
Acronym: TIMEProject
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Laura Marks, Principal Investigator, Florida State University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: STUDY00004768; 5K23AA030602 (NIH)
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Healthy Participants; Feasibility Studies; Acceptability

STUDY DESIGN:
Intervention Model Description: The study is a pilot micro-randomized trial where participants are micro-randomized daily in a 28-day trial to receive different types of messages (episodic-future thinking, reciprocity, or no text message) and enticed by a gaming app to examine the feasibility and acceptability of these strategies to engage participants in a mindfulness mobile health application.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reciprocity (Other): Reciprocity text messages include giving participants a message with an solicited reward (e.g., credits in gaming app, $1).
  Interventions: Other: Mindfulness Smartphone Application
- Episodic Future Thinking (Other): Episodic Future Thinking text messages include giving participants a message that encourages them to think vividly about their future
  Interventions: Other: Mindfulness Smartphone Application
- No text message (Other): Participants receive no text message in this arm
  Interventions: Other: Mindfulness Smartphone Application

INTERVENTIONS:
Other: Mindfulness Smartphone Application — A mindfulness mobile health smartphone application that has mindfulness information and practice videos.

SUMMARY:
The goal of this clinical trial is to examine the feasibility and acceptability of different types of text messages and a integrated gaming app to increase engagement in a mindfulness mobile health application.

1. Does receiving text messages increase engagement in a mindfulness app?
2. Does an integrated gaming app increase engagement in a mindfulness app?

Researchers will examine whether participants engage more in a mindfulness mobile health application if they receive text messages and if they engage in additional gaming app on their smartphone. Participants will:

1. Use a mindfulness and gaming mobile health application for 28-days.
2. Complete a pre-study survey, post-study survey, follow-up interview, and 3-month follow-up survey in addition to daily brief surveys.

DETAILED DESCRIPTION:
Participants who are eligible to participate in the pilot micro-randomized trial (MRT) will be screened and onboarded via Zoom. They will be given baseline measures and trained on using the mindfulness app with integrated gaming app on their smartphone. Micro-randomizations will be used to address scientific questions related to the delivery and personalization of episodic future thinking and reciprocity engagement strategies in addition to gamification across the 28-day trial. The proposed pilot MRT will micro-randomize participants in the morning into one of three options: (i) episodic future thinking text-based prompts, (ii) reciprocity text-based prompts, or (iii) no prompts with equal probability. Participants will receive mobile-based ecological momentary assessments in the evening. EMA data will be paired with usage data from the mindfulness app (e.g., time spent in app, number of sessions, completion of mindfulness videos) to assess the conditions under which participants are receptive to engagement strategies. After 28 days, a follow-up survey questionnaire will be administered and an individual interview will be conducted with each participant. A 3-month follow-up survey will also be administered to participants who complete the study. Our primary outcome in engagement in the mindfulness app, and our secondary outcomes are stress and alcohol use.

ELIGIBILITY:
Inclusion Criteria:

* US-born
* Black
* biological man
* undergraduate college student
* criteria for binge drinking (5 drinks in about 2 hours) or heavy drinking (more than 14 drinks per week).

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Mobile Health Engagement | 1 month
  We will assess engagement in our mindfulness mobile health application by measuring paradata (i.e., time spent in the app, whether or not the app was opened, which content was viewed in the app).

SECONDARY OUTCOMES:
Change in Alcohol Use | Baseline; 1 month; 3 months
  Participants will utilize recall and report the total number of days they consumed alcohol over the last 30 day period
Change in Stress | Baseline; 1 month; 3 months
  Perceived Stress Scale is a 10 question Likert Scale that utilizes a 0-4 range ( 0=no stress and 4=the worst stress ever). With Score Ranges possible from 0-40 that assess the participants perceived stress over the last 30days.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Reid Marks, PhD, Principal Investigator — Florida State University
Locations (1):
- Florida State University Center for Translational Behavioral Science, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided